CLINICAL TRIAL: NCT01958164
Title: A Multicenter, Open-label, Randomised, Clinical Trial to Compare the Efficacy and Safety of Actilyse 2 mg/ 2 ml Versus Saline Solution in Restoring Function of an Occluded Central Venous Access Device
Brief Title: Efficacy and Safety of Actilyse 2 mg/ 2 ml in Comparison to Saline Solution in Patients With Central Venous Access Device Occlusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 135.323
Record Dates: First submitted 2013-10-01; First posted 2013-10-09 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Catheter Obstruction; Vascular Access Devices
MeSH Terms: interventions — Tissue Plasminogen Activator; Saline Solution

ARMS (2):
- Actilyse 2 mg/2 ml (Experimental): First dose of Actilyse 2mg/2ml will be given at time 0. Second dose will be given at 120 if CVAD function has not been restored.
  Interventions: Drug: Actilyse
- Saline solution (NaCl 0.9%) (Sham Comparator): Saline solution will be given at time 0. First dose of Actilyse 2mg/2ml will be given to patients if CVAD function has not been restored.
  Interventions: Drug: Actilyse; Drug: Saline solution

INTERVENTIONS:
Drug: Actilyse — Actilyse 2mg/2ml will be given if the CVAD has not been restored at time 120min.
  Arms: Saline solution (NaCl 0.9%)
Drug: Saline solution — Instil Saline solution 2 ml into the disfunctional CVAD once at time O only for patients enrolled in Group II
  Arms: Saline solution (NaCl 0.9%)
Drug: Actilyse — Instil Actilyse 2 mg/ 2 ml into the dysfunctional CVAD at time O.
  Arms: Actilyse 2 mg/2 ml
Drug: Actilyse — Second dose of Actilyse 2mg/2ml will be given if CVAD has not been restored at time 120min.
  Arms: Actilyse 2 mg/2 ml

SUMMARY:
This is a multicentre, open-label, randomised, phase III study designed to evaluate the efficacy and safety of Actilyse 2 mg/2 ml in the restoration of function of CVAD

ELIGIBILITY:
Inclusion criteria:

* Male and female patients between 18 and 80 years, who signed a written informed consent
* Patients with central venous access device occlusion, which occurred within 24-h before randomisation, where central venous access device is indicated for any of the following: fluid maintenance, chemotherapy, intravenous feeding, haemodialysis, long-term administration of antibiotics or other medication
* Patients with central venous access device occlusion occurred within 24-h before randomisation. Central venous access device is defined by inability to withdraw at least 3 ml of blood from the central venous access device. If multiple lumens are occluded, investigators are to choose and treat only one lumen for the study.
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice and the local legislation. Acceptable level of the following laboratory parameters:

  * hemoglobin ≥ 80 g/L;
  * total white blood cell count ≥ 2.0 x109/L;
  * platelets ≥ 50.0 x109/L;
  * fibrinogen ≥0.5 x lower limit of normal;
  * international normalized ratio <2 x upper limit of normal;
  * activated partial thromboplastin time <2 x upper limit of normal;
  * total protein ≥ 35 g/l;
  * alanine transaminase <20 x upper limit of normal;
  * aspartate transaminase <20 x upper limit of normal;
  * total bilirubin <10 x upper limit of normal;
  * creatinine <6 x upper limit of normal;
  * glucose > 2.8 mmol/l.

Exclusion criteria:

* Any clinical evidence of mechanical or non-thrombotic occlusion
* High risk for bleeding events
* High risk for embolic complications
* Any condition for which bleeding constitutes a significant hazard or would be particularly difficult to manage
* Administration of any fibrinolytic agent within 48 hours before start of study treatment
* Patients who have had any of the following within the previous 48 hours before start of study treatment:

  * surgery
  * obstetrical delivery
  * percutaneous biopsy of viscera or deep tissues
  * puncture of non-compressible vessels
  * active internal bleeding
* Patients who have thrombocytopenia, other hemostatic defects (including those secondary to severe hepatic or renal disease).
* Pregnancy and lactation.
* Previously known positive results from infectious serology for Human Immunodeficiency Virus (HIV) or hepatitis B surface antigen (HBsAg), or hepatitis C virus.
* Known hypersensitivity to alteplase or gentamicin, or any excipient of Actilyse - Body weight <30 kg.
* Administration of any fibrinolytic agent within 48 hours before start of study treatment.
* Participation in another investigational trial within 30 days prior to the Screening Visit.
* Concomitant treatment with angiotensin-converting-enzyme inhibitors.
* Impossibility to infuse fluids at the volume necessary to infuse study drug (2 ml) into the central venous access device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Russia (5):
  - 135.323.1 Boehringer Ingelheim Investigational Site, Akhangelsk
  - 135.323.2 Boehringer Ingelheim Investigational Site, Krasnodar
  - 135.323.3 Boehringer Ingelheim Investigational Site, Krasnoyarsk
  - 135.323.7 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 135.323.5 Boehringer Ingelheim Investigational Site, Samara

RESULTS

PARTICIPANT FLOW:
Groups:
- Actilyse: Patients received one dose of Actilyse 2mg/2ml, administered intravenously, at time 0. A second dose was administered at 120 minutes if central venous access device (CVAD) function had not been restored.
- Saline Solution + Actilyse: Patients received one dose of saline solution (NaCl 0.9% - 2ml), administered intravenously, at time 0. A first dose of Actilyse 2mg/2ml was administered intravenously to patients at 120 minutes if central venous access device (CVAD) function had not been restored.
Period: Overall Study
Arm/Group | Actilyse | Saline Solution + Actilyse
Started | 6 (Randomised and treated) | 10 (Randomised and treated)
Completed | 4 | 5
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomised patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Actilyse | Saline Solution + Actilyse | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Continuous [Mean (Full Range); unit: years] | 56.0 [26 to 74] | 63.9 [35 to 76] | 60.9 [26 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Restored CVAD Function at 120 Min After Administration of the First Dose of Study Medication
Description: Proportion (percentage) of patients with restored central venous access device (CVAD) function at 120 min after administration of the first dose of study medication (i.e. Actilyse® or saline solution).
Time Frame: 120 minutes after first drug administration
Population: Full analysis set (FAS) which included all randomised patients who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Actilyse | Saline Solution + Actilyse
Number analyzed (Participants) | 6 | 10
percentage of participants | 83.3 [35.8 to 99.6] | 10.0 [0.2 to 44.5]
Statistical Analysis 1: Comparison: Actilyse vs Saline Solution + Actilyse; Test type: Superiority or Other; Mean Difference (Net) = 73.3, 95% CI 2-sided [23.3 to 89.3] — Difference calculated as actilyse minus saline solution

2. Secondary Outcome: Restored CVAD Function 30 Minutes After Administration of Study Medication at Time 0
Description: Percentage of patients with restored CVAD function 30 minutes after administration of study medication at time 0 (i.e. Actilyse® or saline solution)
Time Frame: 30 minutes after first drug administration
Population: Full analysis set (FAS) which included all randomised patients who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Actilyse | Saline Solution + Actilyse
Number analyzed (Participants) | 6 | 10
percentage of participants | 66.7 [22.3 to 95.7] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Actilyse vs Saline Solution + Actilyse; Test type: Superiority or Other; Mean Difference (Net) = 66.7, 95% CI 2-sided [20.7 to 90.3] — Difference calculated as actilyse minus saline solution

3. Secondary Outcome: Restored CVAD Function 30 Minutes After Administration of the Second Dose of Study Medication Actilyse
Description: Percentage of patients with restored CVAD function 30 minutes after administration of the second dose of study medication Actilyse (150 minutes after time 0)
Time Frame: 150 minutes after first drug administration
Population: All patients in the FAS who did not have restored CVAD function 120 minutes after first drug administration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Actilyse | Saline Solution + Actilyse
Number analyzed (Participants) | 1 | 9
percentage of participants | 100.0 [2.5 to 100.0] | 55.6 [21.2 to 86.3]

4. Secondary Outcome: Restored CVAD Function 120 Minutes After Administration of the Second Dose of Study Medication Actilyse
Description: Percentage of patients with restored CVAD function 120 minutes after administration of the second dose of study medication Actilyse (240 minutes after time 0)
Time Frame: 240 minutes after first drug administration
Population: All patients in the FAS who did not have restored CVAD function 120 minutes after first drug administration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Actilyse | Saline Solution + Actilyse
Number analyzed (Participants) | 1 | 9
percentage of participants | 100.0 [2.5 to 100.0] | 77.8 [39.9 to 97.2]

5. Secondary Outcome: Percentage of Participants Who Achieved Restored CVAD Function After 1 Dose and 2 Doses, in Patients From the Actilyse Treatment Group.
Description: This endpoint was defined as the number of doses required to achieve restored CVAD function in patients from the actilyse treatment group but was analysed as the percentage of participants who achieved restored CVAD function after 1 dose and 2 doses, in patients from the actilyse treatment group.
Time Frame: 0 minutes and 240 minutes
Population: All patients in the FAS who were randomised to the Actilyse treatment group
Measure: Number; unit: percentage of participants
Arm/Group | Actilyse
Number analyzed (Participants) | 6
percentage of participants
  After 1 dose of Actilyse | 83.3
  After 2 doses of Actilyse | 16.7

ADVERSE EVENTS:
Time Frame: From drug administration until the end of that day
Arm/Group | Actilyse | Saline Solution + Actilyse
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Actilyse (N=6) | Saline Solution + Actilyse (N=10)
Arterial hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was stopped prematurely due to slow recruitment of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.